CLINICAL TRIAL: NCT06796946
Title: Intervention for Antidepressant Deprescription in Primary Care: a Randomized Community Clinical Trial
Brief Title: Deprescription of Antidepressants in Primary Care (DAPriCare)
Acronym: DAPriCare
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Huelva (Other)
Responsible Party: Principal Investigator, Juan Gómez-Salgado, Professor Juan Gómez-Salgado, University of Huelva
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2024-TFG-DEPRES; 2024-TFG-DEPRES (Registry Identifier: Provincial Research Ethics Committee of Cadiz on 07/25/2024 (Spain))
Record Dates: First submitted 2025-01-03; First posted 2025-01-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Deprescription; Antidepressants
Keywords: Deprescribing; antidepressants; primary care; clinical trials; mental health; adverse effects
MeSH Terms: conditions — Psychological Well-Being | interventions — Fluoxetine; Citalopram; Sertraline; Paroxetine; Escitalopram

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Deprescription Partial (Experimental): Deprescription
  Interventions: Drug: Deprescription of Antidepressants (fluoxetine, citalopram, sertraline, paroxetine, and escitalopram)
- No Deprescription (No Intervention): No Deprescription
- Deprescription Total (Experimental)
  Interventions: Drug: Deprescription of Antidepressants (fluoxetine, citalopram, sertraline, paroxetine, and escitalopram)

INTERVENTIONS:
Drug: Deprescription of Antidepressants (fluoxetine, citalopram, sertraline, paroxetine, and escitalopram) — Deprescription of Antidepressants Reduction or elimination of the dose of antidepressants (fluoxetine, citalopram, sertraline, paroxetine, and escitalopram) taken by patients
  Arms: Deprescription Partial; Deprescription Total

SUMMARY:
Introduction The consumption of antidepressants has increased considerably worldwide, including in Spain. Despite their effectiveness in cases of moderate to severe depression, their long-term use in mild cases is questioned. This study aims to evaluate the effectiveness of a deprescribing intervention in primary care, to reduce the unnecessary consumption of these drugs and improve patients' quality of life.

Material and Methods A community-based clinical trial will be carried out before and after in an adult population of residents of an urban area of Cadiz (Spain) who have been prescribed antidepressants in the last year. Participants will be randomly selected and followed up for a predetermined period after consensus.

The intervention will consist of a comprehensive evaluation of antidepressant treatment by a team of health professionals. Factors such as indication, dose, and response to treatment will be evaluated, and the Hamilton scale for anxiety and the Beck Inventory for depression will be used. In those cases where it is considered appropriate, a gradual reduction or suspension of the drug will be proposed, always under medical supervision.

Conclusions This research will contribute to generating scientific evidence on the safety and efficacy of deprescribing in primary care, promoting a more rational use of antidepressants, and improving the quality of life of patients. The results obtained could have important implications for clinical practice and for the development of clinical practice guidelines.

DETAILED DESCRIPTION:
MATERIAL AND METHODS Study design A randomized community clinical trial will be conducted. Population and sample The study population comes from an urban area of Cádiz, in the autonomous community of Andalusia (Spain), with a population profile characteristic of urban areas with access to primary health services. The study sample will include patients of both sexes treated in primary care in the urban area of La Laguna, Cádiz, who meet the following inclusion criteria: being of legal age (≥18 years), having received at least one prescription for an antidepressant in the year before the start of the study and having the physical capacity to go to the health center and the mental capacity to give informed consent. Patients who are minors, have changed health centers, have physical or mental disabilities (including advanced dementia, severe cognitive deficit, advanced Alzheimer's disease, and disability >70%), or are hospitalized at the time of selection are excluded. For the calculation of the sample size, the 325 antidepressant users identified in 2023 in the same primary care area were taken as a reference. Considering the expected effect of the intervention of 10% total or partial deprescription of antidepressants, a precision of 5%, and a confidence interval of 95%, a minimum sample of 98 patients was estimated to achieve clinical significance. An additional 10% was adjusted to this calculation to cover possible losses or refusals to participate in the study, resulting in a final sample of 108 patients. The selection of participants was carried out by simple random sampling, ensuring that all patients in the reference population have the same probability of being chosen, which guarantees a representative sample.

Sampling procedure Data collection will be carried out by accessing the information sources provided by the pharmacy unit of the District of Cádiz, Bahía-La Janda. In this unit, a pseudo-anonymized list of patients who have picked up antidepressants in pharmacies during the year before the start of the study will be obtained, using a mathematical coding system to preserve confidentiality.

The sample will be selected from the pseudo-anonymized list using simple random sampling. Subsequently, the list of selected patients will be sent to the address of the clinical management unit where the study will be conducted, which will be forwarded to the research team. The principal investigator will contact the selected subjects by telephone to invite them to participate in the study.

Intervention The intervention will begin with a first visit (V0), in which each participant will be provided with detailed information about the study and will be asked to sign the informed consent. In this initial visit, relevant variables will be collected through a specific questionnaire, including universal variables, sociodemographic variables, comorbidities, and possible drug interactions. In addition, questionnaires for the evaluation of anxiety and depression symptoms will be administered, such as the Hamilton scale for anxiety and the Beck Inventory for depression.

The intervention process will then consist of a series of visits scheduled in the work diary of the family doctor in charge of the deprescription. In the second visit (V1), the diagnosis and symptoms will be re-evaluated, including the detection of possible interactions or adverse reactions. If adverse effects are identified, the corresponding notification procedure will be followed and the dose will be adjusted if necessary. In a third visit (V2), a telephone follow-up will be carried out, which will include psychotherapeutic reinforcement, and in the final face-to-face visit (V3), the deprescription intervention will continue and the results will be evaluated (Figure 1).

The duration of this sequence of visits will not exceed 60 days from the beginning of the process, and in the final visit, participants will be asked to complete the anxiety and depression questionnaires again.

Outcome Measures and Study Variables Main outcome measures include partial or complete deprescription of antidepressants in participants, which will be quantified to determine the success of the intervention in reducing unnecessary or inappropriate prescribing of these drugs. In addition, the percentage of patients who failed to deprescribe due to withdrawal symptoms, as well as the percentage of patients who refused deprescription, will be recorded to identify barriers to the process.

Other key outcomes include changes in anxiety and depression symptomatology, as measured by the Hamilton Anxiety Rating Scale and the Beck Depression Inventory, respectively. The Hamilton Anxiety Rating Scale (HAM-A) assesses the severity of anxiety symptoms, including aspects such as anxious mood, somatic tensions, insomnia, and worries. The validated Spanish version of the HAM-A has shown a Cronbach's alpha coefficient greater than 0.80, indicating adequate internal consistency for measuring anxiety. Regarding test-retest reliability, it has also yielded satisfactory results, with correlation coefficients that usually exceed 0.75, which supports its stability in repeated assessments. The Beck Depression Inventory (BDI) is a self-administered scale that measures the severity of depressive symptoms, covering aspects such as mood, hopelessness, negative self-evaluation, and physical symptoms associated with depression. In validation studies in the Spanish population, the BDI has shown high levels of internal consistency, with a Cronbach's alpha that usually exceeds 0.85.

In addition, the study will analyze various independent variables such as age, sex, family situation, employment situation, type of antidepressant, and the number of antidepressants prescribed at the time of the study. The diagnosis that initially justified the prescription of antidepressants, the origin of the prescriber (primary care, psychiatry, others), the presence of comorbidities, and the existence of potential interactions with other medications will also be considered.

Data analysis A univariate descriptive analysis of the variables included in the study will be performed. The presence of outliers will be examined and missing data will be quantified, in addition to analyzing the distribution of each variable. Qualitative variables will be described using frequency tables, percentages, and prevalences, while quantitative variables will be summarized using measures of central tendency (mean and median) and dispersion (standard deviation and range). All descriptive analyses will be performed using SPSS software, version 29.

Inferential analyses will then be used to identify relationships between the independent variables and the main outcome variable, which is the total or partial deprescription of antidepressants. Bivariate analyses will be performed to assess possible associations, after studying the normality of the sample using the Kolmogorov-Smirnov test, which will allow the selection of the relevant contrast statistic. If the variables meet the requirements, a multivariate binary logistic regression will be applied to analyze the combined effect of the independent variables on deprescription. Likewise, significant differences between the intervention group and the control group will also be studied, for the results evaluated, using contrast statistics such as T-Student or U Mann-Whitney. Ethical considerations This study will be developed following the international ethical recommendations of the Declaration of Helsinki (Fortaleza, 2013), complying with the ethical principles in biomedical research. The study has a favorable report from the Provincial Research Ethics Committee of Cadiz with the code 2024-TFG-DEPRES.

The provisions of Law 14/2007, of July 3, on biomedical research will be observed, in accordance with its seventeenth provision, as well as Law 41/2002, of November 14, basic regulation of patient autonomy and rights and obligations about clinical information and documentation.

In compliance with current regulations, informed consent was requested from all participants who received a detailed information sheet about the study. The processing of the personal data of the participants was carried out following Regulation (EU) 2016/679 of the European Parliament and of the Council on the Protection of Personal Data (General Data Protection Regulation) and Organic Law 3/2018, of December 5, on the Protection of Personal Data and the Guarantee of Digital Rights. In addition, the study followed the regulations of Royal Decree 957/2020, of November 3, which regulates observational studies with medicines for human use, ensuring compliance with legal and ethical provisions throughout the research process.

ELIGIBILITY:
Inclusion Criteria:

* be of legal age (≥18 years),
* have received at least one antidepressant prescription in the year before the start of the study,
* and have the physical capacity to go to the health center and the mental capacity to give informed consent

Exclusion Criteria:

* minors,
* have changed health centers,
* have physical or mental disabilities (including advanced dementia, severe cognitive deficit, advanced Alzheimer's disease, and disability >70%), or,
* are hospitalized at the time of selection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Anxiety | From enrollment to the end of treatment at 8 weeks
  Hamilton Anxiety Rating Scale (HAM-A) The HAM-A consists of 14 items, each aimed at assessing a different aspect of anxiety as experienced by the individual. These items are rated on a scale, with the total score providing an overall measure of the person's anxiety level.
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Depression | From enrollment to the end of treatment at 8 weeks
  Beck Depression Inventory (BDI) 21 items 4 options (0-3)
  Scores 1-10____________________These ups and downs are considered normal 11-16___________________ Mild mood disturbance 17-20___________________Borderline clinical depression 21-30___________________Moderate depression 31-40___________________Severe depression over 40__________________Extreme depression

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio José Madueño-Caro, Cadiz, Cádiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
To publish article in scientific journal
Supporting Information: Study Protocol